CLINICAL TRIAL: NCT00366977
Title: Efficacy and Cost of State Quitline Policies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Department of Human Services, Oregon (Other Government)
Responsible Party: Jeffrey Fellows, PhD, Kaiser Permanente Center for Health Research
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 1 RO1-CA86242-1; 1R01CA086242 (NIH)
Record Dates: First submitted 2006-08-18; First posted 2006-08-22 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Smoking Cessation; Tobacco Use Cessation; Cost-effectiveness
Keywords: Cessation; Smoking; Quitline; Policies; Counseling
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Cessation; Smoking

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Behavioral: Multi-session telephone counseling
Drug: NRT patches

SUMMARY:
State-sponsored anti-tobacco campaigns are motivating large numbers of smokers to seek advice, assistance, and support to make their cessation efforts more successful. Like many states, Oregon has sponsored the implementation of a statewide telephone quitline to provide information, referrals, and cessation support for callers. This study will answer key policy questions about how to most effectively support smokers who call the Oregon Quitline for assistance. The specific aims are to recruit 4,500 callers to participate in a 3 x 2 randomized trial comparing the cost and cost effectiveness of three levels of behavioral intervention. We will also test two different policies on the availability of nicotine patch therapy. Subjects will be interviewed by telephone at 6 and 12 months to assess smoking status, quit attempts, and use of health plan anc community cessation services. Costs will be assessed separately from the perspectives of the patients, health plans, the State (i.e., Oregon Quitline), and society. Cost per quit and cost per year quality-adjusted years of life saved will be calculated from each of these perspectives.

DETAILED DESCRIPTION:
Anti-tobacco media campaigns in many states are motivating large numbers of smokers to seek advice, assistance, and support to make their cessation efforts more successful. Like many other states, Oregon has sponsored the implementation of a statewide telephone quitline to provide information, referrals, and cessation support for callers. Two investigators on this proposal (Hollis and McAfee) have a contract with the State of Oregon to provide the Oregon Quitline (OQL) services. The purpose of the proposed research effort is to collaborate further with State representatives to answer key policy questions about how to most effectively support smokers who call the OQL for assistance.

Our overall aim is to recruit 4,500 callers to the OQL to participate in a 3 x 2 randomized trial to compare the cost and cost effectiveness of three levels of behavioral intervention. We will also test two different policies regarding the availability of nicotine patch therapy. Subjects will be interviewed by telephone at 6 and 12 months to assess smoking status, quit attempts, and use of health plan and community cessation services. Costs will be assessed separately from the perspective of the patients, health plan, the State (i.e., OQL), and society. The specific aims are described below:

1. Compare the efficacy of three policies for supporting OQL callers:

   * Brief counseling with referral to caller's health plan cessation services (standard service);
   * Moderate counseling, referral to health plan, and one follow-up call to reinforce use of health plan services;
   * Moderate counseling, referral, and availability a multi-session telephonic intervention.
2. Compare the efficacy of two policies regarding the provision of nicotine replacement:

   * No offer of nicotine replacement (current policy);
   * An offer of free nicotine replacement patches.
3. Determine the costs and cost per quit of the additional policy interventions relative to usual care (i.e., standard service) from the following perspectives:

   * Societal perspective (total incremental costs per incremental quit);
   * State perspective (incremental cost per quit for OQL services);
   * Health plan perspective (based on differences in use of health plan cessation services);
   * Participant's perspective (based on differences in out-of-pocket expenses).
4. Determine the incremental cost per year-of-life saved for the alternative policies relative to usual care.

ELIGIBILITY:
Inclusion Criteria:

* 18+
* Speak English or Spanish
* Oregon resident
* Smoke 5 or more cigarettes/day
* Planning to quit within 30 days (or quit within in last 7 days)
* Consent to random assignment and follow-up

Exclusion Criteria:

* Health plan benefit includes free multi-session telephone counseling
* Current or planned pregnancy or breast-feeding
* Heart attack within the preceding month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4614 (Actual)
Dates: Start 2000-06; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Participant self-reported 30 day abstinence from any tobacco at 6 and 12 months, assuming intent to treat.

SECONDARY OUTCOMES:
Participant self-reported (at 6 and 12 months) any tobacco use by type
amount used per day
stage of change
number of quit attempts
use of health plan and community cessation resources
intervention total cost, cost per participant, and cost per quit
incremental cost effectiveness ratios for each intervention compared to baseline
patterns of pharmacotherapy use
out-of-pocket expenses for cessation activities.

CONTACTS AND LOCATIONS:
Overall Officials: Jack F. Hollis, PhD, Principal Investigator — Kaiser Permanente Foundation Hospitals/Center for Health Research; Timothy A McAfee, MD, Principal Investigator — Group Health Center for Health Promotion; Michael J Stark, PhD, Principal Investigator — Oregon Health Division/Center for Disease Prevention Epidemiology
Locations (3):
- United States (3):
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - Oregon Health Division/Center for Disease Prevention Epidemiology, Portland, Oregon
  - Free and Clear, Inc., Seattle, Washington

REFERENCES:
- [Background] Aickin M, Gensler H. Adjusting for multiple testing when reporting research results: the Bonferroni vs Holm methods. Am J Public Health. 1996 May;86(5):726-8. doi: 10.2105/ajph.86.5.726. PMID 8629727
- [Background] Centers for Disease Control and Prevention, National Center for Health Statistics. U.S. Decennial Life Tables for 1989-91. Volume II, State Life Tables Number 38, Oregon. May 1998.
- [Background] Curry SJ, Grothaus LC, McAfee T, Pabiniak C. Use and cost effectiveness of smoking-cessation services under four insurance plans in a health maintenance organization. N Engl J Med. 1998 Sep 3;339(10):673-9. doi: 10.1056/NEJM199809033391006. PMID 9725926
- [Background] Curry SJ, McBride C, Grothaus LC, Louie D, Wagner EH. A randomized trial of self-help materials, personalized feedback, and telephone counseling with nonvolunteer smokers. J Consult Clin Psychol. 1995 Dec;63(6):1005-14. doi: 10.1037//0022-006x.63.6.1005. PMID 8543703
- [Background] Davidson M, Epstein M, Burt R, Schaefer C, Whitworth G, McDonald A. Efficacy and safety of an over-the-counter transdermal nicotine patch as an aid for smoking cessation. Arch Fam Med. 1998 Nov-Dec;7(6):569-74. doi: 10.1001/archfami.7.6.569. PMID 9821833
- [Background] Dobson AJ. An Introduction to Generalized Linear Models. London UK. Chapman & Hall, 1994.
- [Background] Drummond MF, Stoddart GL, Torrance GW. Methods for the economic evaluation of health care programmes. New York: Oxford University Press, 1987.
- [Background] Erickson P, Wilson R, Shannon I. Years of healthy life. Healthy People 2000 Stat Notes. 1995 Apr;(7):1-15. doi: 10.1037/e583992012-001. No abstract available. PMID 11762385
- [Background] Fiore MC, Bailey WC, Cohen SJ, et al Smoking Cessation Clinical Practice Guideline. Rockville MD: U.S. Department of Health and Human Services, 1996. (Public Health Service, Agency for Health Care Policy and Research, Publication No 96-0692.)
- [Background] Fiore MC, Kenford SL, Jorenby DE, Wetter DW, Smith SS, Baker TB. Two studies of the clinical effectiveness of the nicotine patch with different counseling treatments. Chest. 1994 Feb;105(2):524-33. doi: 10.1378/chest.105.2.524. PMID 8306757
- [Background] Fiore MC, Novotny TE, Pierce JP, Giovino GA, Hatziandreu EJ, Newcomb PA, Surawicz TS, Davis RM. Methods used to quit smoking in the United States. Do cessation programs help? JAMA. 1990 May 23-30;263(20):2760-5. PMID 2271019
- [Background] Fiscella K, Franks P. Cost-effectiveness of the transdermal nicotine patch as an adjunct to physicians' smoking cessation counseling. JAMA. 1996 Apr 24;275(16):1247-51. PMID 8601956
- [Background] Gold ME, Siegel JE, Russell LB, Milton CW, eds. Cost-Effectiveness in Health and Medicine. New York: Oxford University Press, 1996.
- [Background] Glasgow RE, Mullooly JP, Vogt TM, Stevens VJ, Lichtenstein E, Hollis JF, Lando HA, Severson HH, Pearson KA, Vogt MR. Biochemical validation of smoking status: pros, cons, and data from four low-intensity intervention trials. Addict Behav. 1993 Sep-Oct;18(5):511-27. doi: 10.1016/0306-4603(93)90068-k. PMID 8310871
- [Background] Hays JT, Croghan IT, Schroeder DR, Offord KP, Hurt RD, Wolter TD, Nides MA, Davidson M. Over-the-counter nicotine patch therapy for smoking cessation: results from randomized, double-blind, placebo-controlled, and open label trials. Am J Public Health. 1999 Nov;89(11):1701-7. doi: 10.2105/ajph.89.11.1701. PMID 10553392
- [Background] Hollis JF, Lichtenstein E, Vogt TM, Stevens VJ, Biglan A. Nurse-assisted counseling for smokers in primary care. Ann Intern Med. 1993 Apr 1;118(7):521-5. doi: 10.7326/0003-4819-118-7-199304010-00006. PMID 8442622
- [Background] Hollis JF, Lichtenstein E, Mount K, Vogt TM, Stevens VJ. Nurse-assisted smoking counseling in medical settings: minimizing demands on physicians. Prev Med. 1991 Jul;20(4):497-507. doi: 10.1016/0091-7435(91)90047-8. PMID 1871078
- [Background] Kenford SL, Fiore MC, Jorenby DE, Smith SS, Wetter D, Baker TB. Predicting smoking cessation. Who will quit with and without the nicotine patch. JAMA. 1994 Feb 23;271(8):589-94. doi: 10.1001/jama.271.8.589. PMID 8301790
- [Background] Korberly B. An open label multicenter trial to evaluate and compare the efficacy of Nicotrol 15mg as part of an OTC intervention package or as a prescription as an aid in smoking cessation. Presented at the meeting of the Society for Research on Nicotine and Tobacco, San Diego, CA, 1999.
- [Background] Lando HA, Pirie PL, Roski J, McGovern PG, Schmid LA. Promoting abstinence among relapsed chronic smokers: the effect of telephone support. Am J Public Health. 1996 Dec;86(12):1786-90. doi: 10.2105/ajph.86.12.1786. PMID 9003138
- [Background] Lando HA, Rolnick S, Klevan D, Roski J, Cherney L, Lauger G. Telephone support as an adjunct to transdermal nicotine in smoking cessation. Am J Public Health. 1997 Oct;87(10):1670-4. doi: 10.2105/ajph.87.10.1670. PMID 9357351
- [Background] Leischow SJ, Muramoto ML, Cook GN, Merikle EP, Castellini SM, Otte PS. OTC nicotine patch: Effectiveness alone and with brief physician intervention. American Journal of Health Behavior 1999; 23:61-69.
- [Background] Lichtenstein E, Brown RA. Current trends in the modification of cigarette dependence. In Bellack AS, Hersen M, Kazdin AE (eds.). International Handbook of Behavioral Modification and Therapy. New York: Plenum Press, 1982, 575-611.
- [Background] Lichtenstein E, Hollis J. Patient referral to a smoking cessation program: who follows through? J Fam Pract. 1992 Jun;34(6):739-44. PMID 1593248
- [Background] Lichtenstein E, Hollis JF, Severson HH, Stevens VJ, Vogt TM, Glasgow RE, Andrews JA. Tobacco cessation interventions in health care settings: rationale, model, outcomes. Addict Behav. 1996 Nov-Dec;21(6):709-20. doi: 10.1016/0306-4603(96)00030-5. PMID 8904937
- [Background] Lichtenstein E, Glasgow RE, Lando HA, Ossip-Klein DJ, Boles SM. Telephone counseling for smoking cessation: rationales and meta-analytic review of evidence. Health Educ Res. 1996 Jun;11(2):243-57. doi: 10.1093/her/11.2.243. PMID 10163409
- [Background] Lippiatt BC. Measuring medical cost and life expectancy impacts of changes in cigarette sales. Prev Med. 1990 Sep;19(5):515-32. doi: 10.1016/0091-7435(90)90050-t. PMID 2122438
- [Background] Lipscomb J, Weinstein MC, Torrance GW. Time preference. In: Gold MR, Siegel JE, Russell LB, Weinstein MC, eds. Cost-effectiveness in Health and Medicine, Ch. 7.. New York: Oxford University Press, 1996.
- [Background] Little RJA, Rubin DB. Statistical analysis with missing data. New York: John Wiley & Sons, 1987.
- [Background] Manning WG, Fryback DG, Weinstein MC. Reflecting uncertainty in cost-effectiveness analysis. In: Gold MR, Siegel JE, Russell LB, Weinstein MC, eds. Cost-effectiveness in Health and Medicine, Ch. 8. New York: Oxford University Press, 1996
- [Background] Marlatt GA and Gordon JR (Eds). Relapse Prevenion: Maintenance strategies in the treatment of addictive behaviors. New York: Guilford Press, 1985.
- [Background] McCullagh P, Nelder JA. Generalized Linear Models. London UK: Chapman & Hall, 1986
- [Background] Meenan RT, Stevens VJ, Hornbrook MC, La Chance PA, Glasgow RE, Hollis JF, Lichtenstein E, Vogt TM. Cost-effectiveness of a hospital-based smoking cessation intervention. Med Care. 1998 May;36(5):670-8. doi: 10.1097/00005650-199805000-00007. PMID 9596058
- [Background] Miller WR, Rollnick S. Motivational Interviewing: Preparing People to Change Addictive Behavior. New York: The Guilford Press, 1991.
- [Background] O'Brien BJ, Drummond MF, Labelle RJ, Willan A. In search of power and significance: issues in the design and analysis of stochastic cost-effectiveness studies in health care. Med Care. 1994 Feb;32(2):150-63. doi: 10.1097/00005650-199402000-00006. PMID 8302107
- [Background] Orleans CT, Schoenbach VJ, Wagner EH, Quade D, Salmon MA, Pearson DC, Fiedler J, Porter CQ, Kaplan BH. Self-help quit smoking interventions: effects of self-help materials, social support instructions, and telephone counseling. J Consult Clin Psychol. 1991 Jun;59(3):439-48. doi: 10.1037//0022-006x.59.3.439. PMID 2071729
- [Background] Ossip-Klein DJ, Giovino GA, Megahed N, Black PM, Emont SL, Stiggins J, Shulman E, Moore L. Effects of a smoker's hotline: results of a 10-county self-help trial. J Consult Clin Psychol. 1991 Apr;59(2):325-32. doi: 10.1037//0022-006x.59.2.325. PMID 2030195
- [Background] Patrick DL, Cheadle A, Thompson DC, Diehr P, Koepsell T, Kinne S. The validity of self-reported smoking: a review and meta-analysis. Am J Public Health. 1994 Jul;84(7):1086-93. doi: 10.2105/ajph.84.7.1086. PMID 8017530
- [Background] Platt S, Tannahill A, Watson J, Fraser E. Effectiveness of antismoking telephone helpline: follow up survey. BMJ. 1997 May 10;314(7091):1371-5. doi: 10.1136/bmj.314.7091.1371. PMID 9161308
- [Background] Proschan MA. A multiple comparison procedure for three- and four-armed controlled clinical trials. Stat Med. 1999 Apr 15;18(7):787-98. doi: 10.1002/(sici)1097-0258(19990415)18:73.0.co;2-m. PMID 10327527
- [Background] Rigotti NA, Arnsten JH, McKool KM, Wood-Reid KM, Pasternak RC, Singer DE. Efficacy of a smoking cessation program for hospital patients. Arch Intern Med. 1997 Dec 8-22;157(22):2653-60. PMID 9531235
- [Background] Rollnick S, Heather N, Bell A. Negotiating behaviour change in medical settings: The development of brief motivational interviewing. Journal of Mental Health 1992; 1:25-37.
- [Background] Shiffman S. Efficacy of nicotine gum and patch under OTC and real-world prescription conditions. Presented at the meeting of the Society for Research on Nicotine and Tobacco, San Diego, CA, 1999.
- [Background] Simon JA, Solkowitz SN, Carmody TP, Browner WS. Smoking cessation after surgery. A randomized trial. Arch Intern Med. 1997 Jun 23;157(12):1371-6. PMID 9201012
- [Background] Sonderskov J, Olsen J, Sabroe S, Meillier L, Overvad K. Nicotine patches in smoking cessation: a randomized trial among over-the-counter customers in Denmark. Am J Epidemiol. 1997 Feb 15;145(4):309-18. doi: 10.1093/oxfordjournals.aje.a009107. PMID 9054234
- [Background] Stevens VJ, Glasgow RE, Hollis JF, Lichtenstein E, Vogt TM. A smoking-cessation intervention for hospital patients. Med Care. 1993 Jan;31(1):65-72. doi: 10.1097/00005650-199301000-00005. PMID 8417271
- [Background] Stevens VJ, Severson H, Lichtenstein E, Little SJ, Leben J. Making the most of a teachable moment: a smokeless-tobacco cessation intervention in the dental office. Am J Public Health. 1995 Feb;85(2):231-5. doi: 10.2105/ajph.85.2.231. PMID 7856783
- [Background] Thompson B, Fries E, Hopp HP, Bowen DJ, Croyle RT. The feasibility of a proactive stepped care model for worksite smoking cessation. Health Educ Res. 1995 Dec;10(4):455-465. doi: 10.1093/her/10.4.455. PMID 10159675
- [Background] Thorndike AN, Rigotti NA, Stafford RS, Singer DE. National patterns in the treatment of smokers by physicians. JAMA. 1998 Feb 25;279(8):604-8. doi: 10.1001/jama.279.8.604. PMID 9486755
- [Background] Velicer WF, Prochaska JO, Rossi JS, Snow MG. Assessing outcome in smoking cessation studies. Psychol Bull. 1992 Jan;111(1):23-41. doi: 10.1037/0033-2909.111.1.23. PMID 1539088
- [Background] Wetter DW, Fiore MC, Baker TB, Young TB. Tobacco withdrawal and nicotine replacement influence objective measures of sleep. J Consult Clin Psychol. 1995 Aug;63(4):658-67. doi: 10.1037//0022-006x.63.4.658. PMID 7673544
- [Background] Wetter DW, Fiore MC, Gritz ER, Lando HA, Stitzer ML, Hasselblad V, Baker TB. The Agency for Health Care Policy and Research Smoking Cessation Clinical Practice Guideline. Findings and implications for psychologists. Am Psychol. 1998 Jun;53(6):657-69. doi: 10.1037//0003-066x.53.6.657. PMID 9633266
- [Background] Wetter DW, Fiore MC, Young TB, McClure JB, de Moor CA, Baker TB. Gender differences in response to nicotine replacement therapy: objective and subjective indexes of tobacco withdrawal. Exp Clin Psychopharmacol. 1999 May;7(2):135-44. doi: 10.1037//1064-1297.7.2.135. PMID 10340153
- [Background] Wetter DW, Kenford SL, Smith SS, Fiore MC, Jorenby DE, Baker TB. Gender differences in smoking cessation. J Consult Clin Psychol. 1999 Aug;67(4):555-62. doi: 10.1037//0022-006x.67.4.555. PMID 10450626
- [Background] Wetter DW, Smith SS, Kenford SL, Jorenby DE, Fiore MC, Hurt RD, Offord KP, Baker TB. Smoking outcome expectancies: factor structure, predictive validity, and discriminant validity. J Abnorm Psychol. 1994 Nov;103(4):801-11. doi: 10.1037//0021-843x.103.4.801. PMID 7822583
- [Background] Zhu SH, Stretch V, Balabanis M, Rosbrook B, Sadler G, Pierce JP. Telephone counseling for smoking cessation: effects of single-session and multiple-session interventions. J Consult Clin Psychol. 1996 Feb;64(1):202-11. doi: 10.1037//0022-006x.64.1.202. PMID 8907100